CLINICAL TRIAL: NCT03716973
Title: An Open Label Pilot Study to Investigate the Response to High Density Stimulation With Medtronic Restore Sensor Technology in Patients With Intractable Neuropathic Pain Who Have Not Had Spinal Surgery
Brief Title: A Study to Investigate High-density Spinal Cord Stimulation in Virgin-back Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 011454
Record Dates: First submitted 2018-10-18; First posted 2018-10-23 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Neuropathic Pain
Keywords: spinal cord stimulation; paraesthesia-free
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: Open label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High density programming (Experimental): High density programming of spinal cord stimulator for paraesthesia-free therapy.
  Interventions: Device: High Density Programming

INTERVENTIONS:
Device: High Density Programming — Patients implanted with Medtronic spinal cord stimulator will have high density programming.

SUMMARY:
This study will look into the effectiveness of spinal cord stimulation (SCS) in reducing chronic neuropathic pain in patients who have not had previous spinal surgery. This will be assessed by comparing the Numerical Rating Scale (NRS) questionnaire responses before and after the SCS intervention.

We will also investigate the effect of HD frequency parameters on the improvement of quality of life, sleep and any adverse events following the spinal cord stimulation.

DETAILED DESCRIPTION:
Traditionally, spinal cord stimulation (SCS) has been used for patients with chronic neuropathic pain following back surgery (a condition known as Failed Back Surgery Syndrome (FBSS)). Although the National Institute for Health and Care Excellence (NICE) also recommends SCS for chronic neuropathic pain without previous back surgery, clinical outcome data is much needed in this patient group. Conventionally, patients receiving SCS are provided with tonic stimulation settings (where they feel tingling and paraesthesia); however newer methods include high-density stimulation (HD) that provides higher energy allowing the voltage to be reduced to subthreshold parameters, hence minimizing the tingling and paraesthesia. HD stimulation is widely offered to patients with SCS as part of routine clinical practice, although no known studies have yet investigated HD settings in patients with neuropathic pain without previous spinal surgery. Therefore, the purpose of this study is to determine the effectiveness of HD settings in patients without previous spinal surgery undergoing SCS. 20 patients without previous spinal surgery who are deemed suitable for SCS as part of NICE guidelines 159 pathway will be recruited for the study.

All patients have a trial of SCS where they will be offered HD settings. If successful (>50% improvement in pain scores) they will be offered permanent implant. Those patients whose pain does not improve with HD settings will be further offered conventional tonic stimulation for one more week. Those patients who do not respond to both tonic and HD settings will be excluded and will not have permanent implant. This will also allow us to investigate the patient's preference between the HD neurostimulator settings and conventional tonic settings. We will also investigate the response to these stimulator settings on health related quality of life. Patients will complete quality of life questionnaires at Baseline, 1-month, 3-months and 12-months post-implant.

ELIGIBILITY:
* Male and female patients between 18-75 years of age who have lumbar radiculopathy who have not undergone any spinal surgery.
* Patients with intractable neuropathic pain due to undergo Percutaneous Spinal Cord Stimulation as part of their standard treatment for lumbar neuropathic pain as per NICE HTA guidance 159 at Barts Health NHS Hospitals. The decision would be made by the multidisciplinary team by reviewing the history, MRI scans and patient choice.
* Patients who have given their written informed consent.
* Female patients of childbearing potential must be using adequate contraception (i.e. using oral or IM contraception or an IUCD) and must have a negative urine pregnancy test.

Exclusion Criteria:

* Patients with diabetes or any underlying neurological condition.
* Patients known to have a condition that in the investigator's judgement precludes participation in the study.
* Patients who have received an investigational drug or have used an investigational device in the 30 days preceding study entry.
* Patients unable to comply with the study assessments and to complete the questionnaires.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | Baseline, 1-month, 3-months, 12months
  Investigate the change in reported pain scores (NRS) following percutaneous spinal cord stimulation (SCS) with Restore Sensor in patients with lumbar radiculopathy who have not undergone any spinal surgery ("virgin back").

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Baseline, 1-month, 3-months, 12months
  low back functional outcome tool
Patient's Global Impression of change (PGIC) | Baseline, 1-month, 3-months, 12months
  A standard seven point scale would be used to assess the SCS outcome.
Pain and Sleep Questionnaire _3 (PSQ_3) | Baseline, 1-month, 3-months, 12months
  A three-item index for the assessment of the impact of pain on sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Mehta, MD, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No